CLINICAL TRIAL: NCT04099498
Title: In-person and Online Healthy Eating Promotion Through Self-regulation (HEP-S): Assessing the Efficacy of a Narrative-based Intervention
Brief Title: In-person and Online Healthy Eating Promotion Through Self-regulation (HEP-S)
Acronym: HEP-S
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Minho (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Paula Cristina Soares de Magalhães da Silva Correia, Junior Researcher, University of Minho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POCI-01-0145-FEDER-028302
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Healthy Eating
Keywords: Self-regulation; Healthy eating; Online; Promotion
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Intervention Model Description: A three-armed randomized controlled trial will be conducted and will include: a standard control group, with no intervention; an online-intervention group, with the program for 20-weeks; and an enhanced-online-intervention group, with the program for 20-weeks embedded with gamification strategies throughout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Control group (No Intervention): This group will not partake in the intervention but will be assessed with the same protocol at the same moments.
- Online-Intervention group (Experimental): This group will take part of the 20-week long online intervention to promote healthy eating. The program will be developed to promote self-regulation skills and strategies about healthy eating among elementary school-aged children and each week will include: i) a narrative embedded with self-regulation skills and strategies; ii) a weekly parental involvement activity; and iii) a weekly group synchronous videoconference session with a trained educational psychologist serving as a mediator.
  Interventions: Behavioral: Online Program: Healthy Eating Promotion with Self-regulation
- Enhanced-online-Intervention Group (Experimental): This group will take part of the 20-week long online intervention to promote healthy eating. The program will be developed to promote self-regulation skills and strategies about healthy eating among elementary school-aged children and each week will include: i) a narrative embedded with self-regulation skills and strategies; ii) a weekly parental involvement activity; and iii) a weekly group synchronous videoconference session with a trained educational psychologist serving as a mediator. In addition, gamification strategies (e.g., points for each complete activity, feedback) will be implemented in order to promote engagement with the program and activities.
  Interventions: Behavioral: Enhanced Online Program: Healthy Eating Promotion with Self-regulation

INTERVENTIONS:
Behavioral: Online Program: Healthy Eating Promotion with Self-regulation — Online-Intervention group
  Arms: Online-Intervention group
Behavioral: Enhanced Online Program: Healthy Eating Promotion with Self-regulation — Enhanced-online-Intervention Group
  Arms: Enhanced-online-Intervention Group

SUMMARY:
Obesity has more than doubled worldwide since 1980. The challenge with obesity, as with many other modern diseases, is that the solution may not rely on the medical side of the chain but rather on the individual via modifiable factors and behavioral changes such as eating habits and physical activity.

The main goals of Healthy Eating Promotion with Self-regulation (HEP-S) are to design, implement, and evaluate the efficacy of an online intervention that promotes healthy eating among elementary school children using narratives involving self-regulation themes and skills. Self-regulation (SR) refers to the processes that allow individuals to proactively control the personal, behavioral, and environmental influences that impact their behavior, including eating. The focus of this project is not on delivering knowledge per se about healthy eating but rather on promoting and developing a set of transversal skills and strategies on the healthy habits' domain. We chose this focus because we recognized that beliefs about healthy eating have a stronger influence on eating behavior than factual knowledge about food. At the core of this intervention are the narratives, an important educational tool that favors child development; they allow readers to reflect on themselves and their behavior through the characters presented. Narratives also instigate the debate and the uncovering of different perspectives on how to cope with daily dilemmas. By using stories to initiate discussion and reflection, it is expected that a change of beliefs will occur, thus prompting a behavioral change.

In today's world, there is an increasing need to dematerialise procedures so interventions can reach more people at a lower cost. Thus, it is important to test the feasibility of the online version of the intervention.

Overall, it is expected that children taking part of the intervention will, at the end of the intervention, increase their use of SR strategies for healthy eating, enhance their sense of self-efficacy for healthy eating, and increase their consumption of healthy foods. Additionally, it is expected that their knowledge on the topic will increase, that their food preferences become healthier, and that they will display more positive perceptions and attitudes about the topic. Lastly, it is expected that participants enrolled in the enhanced-online-intervention group will be more engaged in the intervention than the online-intervention group.

DETAILED DESCRIPTION:
HEP-S program is grounded on the Self-regulation (SR) approach, which has several features that make it unique when it comes to health promotion. Grounded on Social Cognitive Theory, SR subsumes the processes that allow individuals to proactively control the personal, behavioural, and environmental influences that impact human behavior, including eating. These processes are intrinsically cyclic and interdependent, open and dynamic, and proceed through three main phases: the preceding phase, the performance or volitional control phase, and the self-reflection phase (or Planning, Execution, and Evaluation). The SR process is under the influence of the individual and can, therefore, be taught and improved. Thus, the agent role of the individual throughout the process is key to become in control and autonomous.

Although individuals may be influenced and regulated by external factors and agents, exclusively relying on external regulation does not allow for the individual to develop adaptive competences and skills, such as choosing a healthy snack. Thus, to self-regulate their behaviour and become increasingly autonomous, individuals must progressively shift from external regulation to a model that supports and provides feedback. SR can be essential in the processes of healthy eating as individuals who SR their behavior are likely to plan and systematically use a set of cognitive and metacognitive strategies to meet self-set goals. Thus, the effective use of SR strategies to achieve one's goal is part of a key process in maintaining an individual's motivation to reach a self-set goal, such as eating healthily.

In several studies, researchers have successfully implemented self-management programs among individuals with various health conditions, such as heart disease, or obesity. With the help of these programs, individuals were able to manage their health conditions and improve their quality of life and wellbeing. Still, these programs focused on health promotion within a disease management context, not on prevention and promotion of a healthy lifestyle. Thus, the current proposal will address this gap by focusing on healthy eating promotion among children.

The HEP-S is a 20-week narrative-based intervention designed to promote healthy eating through the teaching and development of a set of transversal skills and strategies within that domain. The program will be implemented online using the online tool Canvas®. Canvas® is a learning management system that allows, among other things, to create modules of content, attach files, share materials, create discussion forums, and conduct videoconferences. Each child will be provided with a unique login to the Canvas® of the class. The program has two main components: i) the weekly synchronous session, which includes the reading of the chapter, the discussion and reflection about the lessons conveyed in the chapter, and the strengthening of learning through a consolidation activity; and ii) the weekly parental involvement activity, which is conceived to consolidate learning of the SR processes and skills.

At the core of this intervention are the narratives. Narratives, or story-tools, are important educational tools that favor child development. They allow readers to reflect on themselves and their own behaviour through the characters; they instigate the debate and the uncovering of different perspectives of how to cope with every-day dilemmas. Through the characters and plots, these story-tools create opportunities from which the readers can experience and develop autonomous behaviors and promote SR in a given domain (e.g., learning, healthy eating). Extensive extant research has examined and demonstrated the efficacy of using story-tools to promote SR strategies. In this study, excerpts of two narratives will be used as the prompt for, and instigate, discussion and reflection about healthy eating. Specifically, Yellow's Trials and Tribulations, and The Hill of the Bald Trees and Other Stories.

There will be two intervention groups: the online-intervention and enhanced-online-intervention. What differentiates these groups is that the enhanced-online-intervention group counts with the inclusion of gamification strategies within the dynamic of the program. Gamification consists in the use of game design elements in a non-game context. Non-game contexts can be education, health, and business. Examples of game design elements are the narrative context, feedback, reputation, ranks, levels, competition, relational support. Considering the engaging nature of games, it is expected that embedding some of their design and motivational features will contribute to the: i) creation of more engaging and fun contexts or environments; ii) enhancement of the degree and depth of participants' engagement; iii) promotion of learning opportunities; and iv) motivate individuals to engage in the task at hand.

Goals and expected outcomes:

The main purpose of this study is to evaluate the efficacy of an online intervention designed to promote healthy eating by fostering the use of SR strategies among school-aged children. Thus, the major goals are to promote children's use of SR strategies for healthy eating, to strengthen their sense of self-efficacy regarding healthy eating, to increase consumption and knowledge about healthy eating; to contribute to healthier food preferences; and contribute to more positive attitudes and perceptions about healthy eating. Concomitantly, we want to assess the feasibility of conducting an online intervention with this population and examine the advantages of embedding the program with gamification strategies.

Overall, it is expected that children taking part of the intervention will increase their use of SR strategies for healthy eating, enhance their sense of self-efficacy for healthy eating, and increase their consumption of healthy foods. Additionally, it is expected that their knowledge on the topic will increase, and that they will display more positive perceptions and attitudes about the topic. Lastly, it is expected that participants enrolled in the enhanced-online-intervention group will be more engaged in the intervention than the online-intervention group.

Participants:

Children from the 5th and 6th grades will be recruited by first contacting Portuguese elementary and middle schools and inviting them to participate. Orientation sessions will be held at schools for all parents of children in the target grades to explain the project and its rationale, and to invite them to enroll their child. The study will be introduced as a program to promote healthy lifestyles among school-aged children, which aims to monitor relevant engagement variables and examine children's, parents', and teachers' perceptions of the utility and feasibility of these interventions.

Retention and incentives for the participants:

The following strategies will be undertaken to minimize attrition. First, prior to the intervention, the researchers will organize orientation sessions with parents to present the project and explain its pertinence and rationale. Second, parents who agree to let their child participate in the program will sign a participation agreement detailing their responsibility as guarantors of their child's involvement in the program. Third, the registration e-mail for children to log in into the platform will be of their parents, and reminder emails will be sent whenever there is an activity or task available in the platform. Lastly, check-up sessions with parents will be carried mid-through the program.

Informed consent and randomization:

During the orientation session, parents who allow their child to participate in the program will complete the first assessment protocol in loco, as well as complete the informed consent form. In the informed consent, the following aspects will be covered: i) description of the program, accompanied by a timeline; ii) duties of the parents as guarantors of their child's involvement in the program; and iii) what it is expected from them in terms of their involvement with the program and its activities. Genuine randomization at the individual level will not be possible as participants originating from the same class and school will have to be allocated to the same treatment condition to prevent between-group contamination. To address this difficulty, each school that accepts to enroll in the study will be randomly attributed a number associated with one of the conditions (i.e. control, intervention, and enhanced-intervention) in a 1:1:1 basis.

Proposed sample size:

Considering this longitudinal design, the sample size was computed using G*Power software. In the calculation of the sample, we considered a 0.2 effect size, an alpha level of 0.05, a desired statistical power of 0.8, five measures, three research groups (i.e. control, online-intervention, enhanced-online-intervention), and a 20% dropout rate. This analysis suggested that a total of 150 participants will be recruited, with 50 participants per group.

Statistics:

Descriptive analyses will be computed to describe all participants' characteristics. Specifically, we will use chi-square tests and independent t-tests to compare groups on the distributions according to sex, age group, BMI classification and others. To assess the effectiveness of the HEP-S intervention program, we will develop linear mixed-effect models to specifically assess groups differences over time. All analyses will be conducted using SPSS, and p values below .05 will be considered statistically significant.

Blinding and data access:

The assessment protocol will be completed by children and will not be available for parents to consult or to the educational psychologist conducting the sessions. Each child will be attributed a unique code. Moreover, data will be analyzed by an external statistician who will be blind to the treatment conditions of each data set. Lastly, only the principal investigator and the statistician will have access to the full data set.

The standard procedure to conduct studies in the Portuguese school context requires an a priori evaluation and validation of the project by the Ministry of Education and by the Ethics Committee of the University of Minho before researchers can invite schools to participate. Participation in the program is entirely voluntary, and parents and children are informed that their involvement in the school's activities will not be affected by their decision on whether or not to participate. Parents and children are informed they can withdraw from the program at any time. We fully recognize our responsibilities for child protection, so the project will ensure an environment where children feel secure, feel free to either participate or leave the study at any time, are encouraged to talk, and are listened to. In order to work with children, researchers must present their criminal records during the job application. This protocol will be held to meet high ethical standards.

Lastly, the procedures for personal data storage, handling, and protection will comply with the newest General Data Protection Regulation policies. Particularly, to ensure privacy and anonymity, pseudonymisation will be carried out. This is a process that transforms personal data into a data set that cannot be linked to a particular subject unless other piece of information is added (e.g., decryption key). Usually, these data are stored in different locations.

ELIGIBILITY:
Inclusion Criteria:

* Access to a computer equipped with camera and speakers at home;
* Internet access at home;
* Children have to read, speak and write Portuguese fluently;
* Parents have to provide a written consent for their children to participate;
* Children have to provide a written agreement of willingness to participate;
* Parent have to sign the informed consent;
* Parents have to be willing to participate in the parental involvement activities;
* Parents have to have an e-mail account or be willing to create one;

Exclusion Criteria:

* Any acute or chronic condition, or learning disabilities that would limit the ability of the patient to participate in the study
* Refusal to give informed consent

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Socio-demographic Questionnaire. | baseline
  The participants will be asked about their gender, age and grade.
Change of Self-Regulation Processes towards Healthy Eating at 20 weeks from baseline | 20 weeks after baseline
  An adapted version of the Self-Regulation for Health Scale. (Mattos, et. al. 2018) was used to evaluate the self-regulation processes towards healthy eating that participants are guided by. The scale has nine statements regarding the participant's self-regulation towards healthy eating (e.g., I pay attention to information on healthy eating, I apply that knowledge on a daily basis). Responses are scored from 1 (never) to 5 (always) on a Likert-like scale and summed to create a composite score from nine to 45, with higher scores implying more self-regulation.
Change of Self-Regulation Processes towards Healthy Eating at 3 months from the end of the intervention | 3-months after end of the intervention
  An adapted version of the Self-Regulation for Health Scale. (Mattos, et. al. 2018) was used to evaluate the self-regulation processes towards healthy eating that participants are guided by. The scale has nine statements regarding the participant's self-regulation towards healthy eating (e.g., I pay attention to information on healthy eating, I apply that knowledge on a daily basis). Responses are scored from 1 (never) to 5 (always) on a Likert-like scale and summed to create a composite score from nine to 45, with higher scores implying more self-regulation.
Change of Self-Regulation Processes towards Healthy Eating at 6-months after the last assessment | 6-months after the last assessment
  An adapted version of the Self-Regulation for Health Scale. (Mattos, et. al. 2018) was used to evaluate the self-regulation processes towards healthy eating that participants are guided by. The scale has nine statements regarding the participant's self-regulation towards healthy eating (e.g., I pay attention to information on healthy eating, I apply that knowledge on a daily basis). Responses are scored from 1 (never) to 5 (always) on a Likert-like scale and summed to create a composite score from nine to 45, with higher scores implying more self-regulation.
Change of Students' Attitudes and Perceptions on Healthy Eating at 20 weeks from the baseline | 20 weeks after baseline
  An adaptation of the Students' Attitudes and Perceptions on the Health Instrument (Mattos et al., 2018) will be used. This instrument has 17 statements about student's attitudes and perceptions of the importance of healthy eating (e.g., Eating fruit and vegetables will help me growing up). Responses are scored as true or false, and the correct answers will be summed to create a composite score that ranged from 0 to 17, with higher scores implying more positive attitudes through healthy eating.
Change of Students' Attitudes and Perceptions on Healthy Eatingat 3 months from the end of the intervention | 3-months after end of the intervention
  An adaptation of the Students' Attitudes and Perceptions on the Health Instrument (Mattos et al., 2018) will be used. This instrument has 17 statements about student's attitudes and perceptions of the importance of healthy eating (e.g., Eating fruit and vegetables will help me growing up). Responses are scored as true or false, and the correct answers will be summed to create a composite score that ranged from 0 to 17, with higher scores implying more positive attitudes through healthy eating.
Change of Students' Attitudes and Perceptions on Healthy Eating at 6-months after the last assessment | 6-months after the last assessment
  An adaptation of the Students' Attitudes and Perceptions on the Health Instrument (Mattos et al., 2018) will be used. This instrument has 17 statements about student's attitudes and perceptions of the importance of healthy eating (e.g., Eating fruit and vegetables will help me growing up). Responses are scored as true or false, and the correct answers will be summed to create a composite score that ranged from 0 to 17, with higher scores implying more positive attitudes through healthy eating.
Change of Knowledge of Healthy Eating at 20 weeks from the baseline | 20 weeks from the baseline
  This questionnaire was developed to assess school-age children's (six to 17 years old) declarative knowledge about healthy eating (Pereira, et al. 2018). The questionnaire was built by a team comprised by several specialists (psychologists, teachers, medical doctors, and nurses) and the items were based on the directives by the Portuguese General Directorate for Health (DGS, 2017). The questionnaire consists of 15 statements and participants had to rate their agreement regarding each statement (e.g., "our meal should contain varied and colourful foods"; "going to school without having breakfast does not interfere with my school performance"). Responses to individual items were scored from one (totally disagree) to five (totally agree) in a Likert-like format. The alpha of Cronbach was .73. Responses of each participant were summed to create a composite score ranging from 15 to 75, with higher scores implying more knowledge of healthy eating.
Change od Knowledge of Healthy Eating at 3 months from the end of the intervention | 3-months after end of the intervention
  This questionnaire was developed to assess school-age children's (six to 17 years old) declarative knowledge about healthy eating (Pereira, et al. 2018). The questionnaire was built by a team comprised by several specialists (psychologists, teachers, medical doctors, and nurses) and the items were based on the directives by the Portuguese General Directorate for Health (DGS, 2017). The questionnaire consists of 15 statements and participants had to rate their agreement regarding each statement (e.g., "our meal should contain varied and colourful foods"; "going to school without having breakfast does not interfere with my school performance"). Responses to individual items were scored from one (totally disagree) to five (totally agree) in a Likert-like format. The alpha of Cronbach was .73. Responses of each participant were summed to create a composite score ranging from 15 to 75, with higher scores implying more knowledge of healthy eating.
Change of Knowledge of Healthy Eating at 6-months after the last assessment | 6-months after the last assessment
  This questionnaire was developed to assess school-age children's (six to 17 years old) declarative knowledge about healthy eating (Pereira, et al. 2018). The questionnaire was built by a team comprised by several specialists (psychologists, teachers, medical doctors, and nurses) and the items were based on the directives by the Portuguese General Directorate for Health (DGS, 2017). The questionnaire consists of 15 statements and participants had to rate their agreement regarding each statement (e.g., "our meal should contain varied and colourful foods"; "going to school without having breakfast does not interfere with my school performance"). Responses to individual items were scored from one (totally disagree) to five (totally agree) in a Likert-like format. The alpha of Cronbach was .73. Responses of each participant were summed to create a composite score ranging from 15 to 75, with higher scores implying more knowledge of healthy eating.
Change of Self-Efficacy to Regulate Eating Habits for Children at 20 weeks from the baseline | 20 weeks after baseline
  We will use an adaptation of the questionnaire "Self-Efficacy to Regulate Eating Habits" developed by Bandura (2005) in this project. The measure will assess the perceived capability to regulate and to adopt healthy eating habits in different daily situations (e.g., "While watching television"). This version consists in 15 adapted situations, in which participants will have to respond if they can choose healthy food choices or not in a Likert-like format, scored from one (not capable) to six (capable, for sure).
Change of Self-Efficacy to Regulate Eating Habits for Children at 3 months from the end of the intervention | 3-months after end of the intervention
  We will use an adaptation of the questionnaire "Self-Efficacy to Regulate Eating Habits" developed by Bandura (2005) in this project. The measure will assess the perceived capability to regulate and to adopt healthy eating habits in different daily situations (e.g., "While watching television"). This version consists in 15 adapted situations, in which participants will have to respond if they can choose healthy food choices or not in a Likert-like format, scored from one (not capable) to six (capable, for sure).
Change of Self-Efficacy to Regulate Eating Habits for Children at 6 months after the end of the last assessment | 6 months after the end of the last assessment
  We will use an adaptation of the questionnaire "Self-Efficacy to Regulate Eating Habits" developed by Bandura (2005) in this project. The measure will assess the perceived capability to regulate and to adopt healthy eating habits in different daily situations (e.g., "While watching television"). This version consists in 15 adapted situations, in which participants will have to respond if they can choose healthy food choices or not in a Likert-like format, scored from one (not capable) to six (capable, for sure).
Change of Healthy Eating and Physical Activity Self-Efficacy in children at 20 weeks after baseline | 20 weeks after baseline
  This measure was developed to assess self-efficacy related to enacting healthy eating and activity behaviours in children (Lassetter et al., 2017). An adapted version of the HEPASEQ-C was developed and consists of nine items with response options on a 6-point Likert-type scale, ranging from "There is no way I can do this" to "I believe I can do this". Seven items focus on self-efficacy related to healthy eating. For example, one item says, "I will eat healthy food even when my friends eat food that is not healthy."
Change of Healthy Eating and Physical Activity Self-Efficacy in children at 3 months after the end of the intervention | 3-months after end of the intervention
  This measure was developed to assess self-efficacy related to enacting healthy eating and activity behaviours in children (Lassetter et al., 2017). An adapted version of the HEPASEQ-C was developed and consists of nine items with response options on a 6-point Likert-type scale, ranging from "There is no way I can do this" to "I believe I can do this". Seven items focus on self-efficacy related to healthy eating. For example, one item says, "I will eat healthy food even when my friends eat food that is not healthy."
Change of Healthy Eating and Physical Activity Self-Efficacy in children at 6 months after the end of the last assessment | 6 months after end of the last assessment
  This measure was developed to assess self-efficacy related to enacting healthy eating and activity behaviours in children (Lassetter et al., 2017). An adapted version of the HEPASEQ-C was developed and consists of nine items with response options on a 6-point Likert-type scale, ranging from "There is no way I can do this" to "I believe I can do this". Seven items focus on self-efficacy related to healthy eating. For example, one item says, "I will eat healthy food even when my friends eat food that is not healthy."
Change of the Healthy Eating and Physical Activity Behaviour Recall for Children at 20 weeks after baseline | 20 weeks after baseline
  This measure was developed as a complement to the previous questionnaire and aimed to recall 'children's behaviors in terms of healthy eating and physical activity (Lassetter et al., 2017). The Portuguese version of this questionnaire consists of 9 items, two of which are in an open response format allowing children to write the actual foods they ate. For example, one of these two items states, "The last time I ate a snack at a friend's house, I ate __________." The other seven items include two yes/no items, and the remaining six items had response options that were presented using an ordinal scale.
Change of Healthy Eating and Physical Activity Behaviour Recall for Children at 3-months after end of the intervention | 3-months after end of the intervention
  This measure was developed as a complement to the previous questionnaire and aimed to recall 'children's behaviors in terms of healthy eating and physical activity (Lassetter et al., 2017). The Portuguese version of this questionnaire consists of 9 items, two of which are in an open response format allowing children to write the actual foods they ate. For example, one of these two items states, "The last time I ate a snack at a friend's house, I ate __________." The other seven items include two yes/no items, and the remaining six items had response options that were presented using an ordinal scale.
Change of Healthy Eating and Physical Activity Behaviour Recall for Children at 6 months after end of the last assessment | 6 months after end of the last assessment
  This measure was developed as a complement to the previous questionnaire and aimed to recall 'children's behaviors in terms of healthy eating and physical activity (Lassetter et al., 2017). The Portuguese version of this questionnaire consists of 9 items, two of which are in an open response format allowing children to write the actual foods they ate. For example, one of these two items states, "The last time I ate a snack at a friend's house, I ate __________." The other seven items include two yes/no items, and the remaining six items had response options that were presented using an ordinal scale.

SECONDARY OUTCOMES:
Weekly Diary | 20 weeks
  Each child will use a weekly diary to set goals, plan activities, and monitor his or her own performance. This will allow monitoring the individual progress of children in the program and, simultaneously, to create another moment to reflect about, and consolidate, the learning acquired in the program. Questions will invite children to reflect on what they have learn with the narrative, the synchronous session, and the parental involvement activity of that week. Additionally, questions regarding participants' engagement in the program that week will also be included. Lastly, concrete questions about their food intake will also be covered in the weekly journal.
Satisfaction Questionnaire | 20 Weeks after the baseline
  The research team will develop a satisfaction questionnaire based on previous satisfaction instruments used with this population. The questionnaire will address aspects of utility and feasibility of the program and perceived support by the educational psychologist from the students' perspective.
Engagement Assessment | 20 weeks
  Engagement in the program will be assessed through the analysis of the interactions of children in the online platform. Examples include number of activities completed, comments to peers' posts.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Magalhaes, PhD, Principal Investigator — Psychology Research Cente r (CIPsi) of University of Minho
Locations (1):
- School of Psychology, University of Minho, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Zimmerman BJ. Self-Efficacy: An Essential Motive to Learn. Contemp Educ Psychol. 2000 Jan;25(1):82-91. doi: 10.1006/ceps.1999.1016. PMID 10620383
- [Background] Clark NM, Zimmerman BJ. A social cognitive view of self-regulated learning about health. Health Educ Behav. 2014 Oct;41(5):485-91. doi: 10.1177/1090198114547512. PMID 25270173
- [Background] Rosario P, Mourao R, Nunez JC, Gonzalez-Pienda J, Solano P, Valle A. [Evaluating the efficacy of a program to enhance college students' self-regulation learning processes and learning strategies]. Psicothema. 2007 Aug;19(3):422-7. Spanish. PMID 17617980
- [Derived] Magalhaes P, Silva C, Pereira B, Figueiredo G, Guimaraes A, Pereira A, Rosario P. An online-based intervention to promote healthy eating through self-regulation among children: study protocol for a randomized controlled trial. Trials. 2020 Sep 14;21(1):786. doi: 10.1186/s13063-020-04685-5. PMID 32928277